CLINICAL TRIAL: NCT05442372
Title: Prevalence of Hepatitis B Virus Infection in Pregnancy
Brief Title: Prevalence of HBV in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Maher, Lecturer of Tropical Medicine and Gastroenterology, Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Hepatitis B in pregnancy
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Pregnancy; Prevalence
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The most common mode of HBV transmission is materno-fetal transmission mainly during labor. This study aims to estimate the seroprevalence of HBV infection and the possible risk factors of HBV acquisition in pregnant women in Upper Egypt and to evaluate the predictive value of HBeAg and quantitative HBsAg as surrogate markers for high viremia in pregnant women.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a cause of a vaccine-preventable life-threatening infection of the liver. Worldwide, the estimated number of cases of chronic HBV infection is 296 million cases with about 820 000 deaths, mostly due to liver cirrhosis and hepatocellular carcinoma. The prevalence of HBV infection among pregnant women is estimated to be 1.5-9.5%. The most important risk factor of materno-fetal transmission is high viremia. Other factors include hepatitis B e antigen (HBeAg) seropositivity, HBV S variant, and threatened preterm labor. Quantitative hepatitis B surface antigen (HBsAg) was postulated as a surrogate marker for HBV high viremia in pregnant women by many authors. This study aims to estimate the seroprevalence of HBV infection and the possible risk factors of HBV acquisition in pregnant women in Upper Egypt and to evaluate the predictive value of HBeAg and quantitative HBsAg as surrogate markers for high viremia in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women

Exclusion Criteria:

-

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pregnant women attending antenatal care clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
HBsAg | 6 months
  HBsAg prevalence in pregnancy
Risk factors of HBV in pregnancy | 6 months
  Operations, blood transfusion, dental procedures, tattooing, family history of HBV

SECONDARY OUTCOMES:
correlation between HBeAg and quantitative HBsAg with viral load | 6 months
  to evaluate the predictive value of HBeAg and quantitative HBsAGg as surogate markers for high viraemia in pregnant women hbe ag

CONTACTS AND LOCATIONS:
Overall Officials: Amira Maher, MD, Principal Investigator — Faculty of Medicine, Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt